CLINICAL TRIAL: NCT05716061
Title: Comparison of Median, Intermediate and Lateral Approach to Sacral Erector Spinae Plane Block: a Cadaveric and Radiologic Study
Brief Title: A Cadaveric and Radiologic Study of Sacral Erector Spinae Plane Block (ESPB)
Acronym: ESPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Collaborators: Karadeniz Technical University (Other); Ankara University (Other)
Responsible Party: Principal Investigator, Bilge Olgun Keles, Assistant professor, Giresun University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/229 -13
Record Dates: First submitted 2023-01-21; First posted 2023-02-08 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Nerve Block
Keywords: cadaver study; erector spinae plane block; anatomic dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- median approach (Experimental): Sacral ESPB performed from the median sacral crest of 2.level of sacrum.
  Interventions: Procedure: Sacral ESPB
- intermediate approach (Active Comparator): Sacral ESPB performed bilateral and between the median and intermediate sacral crest of 2.level of sacrum.
  Interventions: Procedure: Sacral ESPB

INTERVENTIONS:
Procedure: Sacral ESPB — Cadaver study

SUMMARY:
The goal of this cadaveric study is to learn about the distribution of contrast agent in ultrasound-guided sacral ESPB. The main questions it aims to answer are

1. Which nerves are affected by this block.
2. Which approach is the best for optimal analgesia in human

DETAILED DESCRIPTION:
4 embalmed cadavers will be divided into groups of 2 and sacral ESPB will be made with 2 different methods. The cadavers will be removed from the solution 48 hours before and will be placed in the prone position, there will be no history of trauma or surgery in the sacral region of the cadavers, and no dissection will be performed from the sacral regions.

In the median approach, the probe will be placed on the cadaver, which was previously placed in the prone position, using a 12-18 megahertz high-frequency linear probe with ultrasound to form a right angle to the sacral crest. After being placed parallel to the sacrum and observing the median crest, a 50 mm echogenic needle will be inserted by advancing the implant towards the second sacral level. After touching the crest, the distribution will be observed by retreating 1mm and making 1 cc of serum physiologic. Then all 40 ml of methylene blue and radiocontrast solution will be given. In the intermediate approach; From the second sacral level, 20 ml of red acrylic dye and a solution containing radiocontrast will be given to the right and left by entering the sulcus between the median and intermedian crests with the same technique, using the same technique, under the guidance of ultrasound. After the procedure, sacral tomography will be performed on the cadavers. The spread of radiocontrast material will be observed and their reconstruction will be performed. Later, anatomical dissection will be performed on the cadavers and the spread of the dyes given will be observed. Which of the sacral intervention methods is more effective in clinical practice will be evaluated.

Estimated durations of the study;

1. Removing the cadavers from the solution 48 hours before, performing the block, going to the radiology and performing the CT scan, coming to the anatomy laboratory and performing the dissection: 3 days
2. Reconstruction and interpretation of radiology images: 1 week
3. Interpretation of anatomical dissection: 1 week
4. Evaluation and writing of the study: 1 month

ELIGIBILITY:
Inclusion Criteria:

* Embalmed cadaver

Exclusion Criteria:

* None of the cadavers had a history of trauma or surgery in the sacral region

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-18 (Actual)

PRIMARY OUTCOMES:
Completion of blocks for 4 cadavers | 3 days
  Ultrasound guided sacral ESPB will be performed on 4 cadavers in 2 different approaches
Completion of computed tomography of 4 cadavers | 3 day
  Computed tomography will be taken in 4 cadavers to observe the distribution of the radiocontrast material given to 2 different regions.

SECONDARY OUTCOMES:
Completion of dissection of 4 cadavers | 3 days
  Four cadaveric specimens will be dissected in order to detect dye spread through tissue compartments

CONTACTS AND LOCATIONS:
Overall Officials: Necati Salman, Study Chair — Ankara University; Selami İnce, Study Chair — Beytepe Hospital; Elvan Tekir Yılmaz, Study Chair — Giresun University; Habip Birinci, Study Chair — Giresun University; Ali Faruk Özyaşar, Study Chair — Karadeniz Technical University; Aysun Uz, Study Chair — Ankara University
Locations (1):
- Bilge Olgun Keleş, Giresun, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tulgar S, Senturk O, Thomas DT, Deveci U, Ozer Z. A new technique for sensory blockage of posterior branches of sacral nerves: Ultrasound guided sacral erector spinae plane block. J Clin Anesth. 2019 Nov;57:129-130. doi: 10.1016/j.jclinane.2019.04.014. Epub 2019 Apr 15. No abstract available. PMID 30999197
- [Result] Aksu C, Gurkan Y. Sacral Erector Spinae Plane Block with longitudinal midline approach: Could it be the new era for pediatric postoperative analgesia? J Clin Anesth. 2020 Feb;59:38-39. doi: 10.1016/j.jclinane.2019.06.007. Epub 2019 Jun 13. No abstract available. PMID 31203111
- [Result] Hamilton DL. The erector spinae plane block: Time for clarity over anatomical nomenclature. J Clin Anesth. 2020 Jun;62:109699. doi: 10.1016/j.jclinane.2020.109699. Epub 2020 Jan 11. No abstract available. PMID 31935572
- [Result] Nanda M, Allan JD, Rojas A, Steele PJ, McMillan DT, Park J, Arora H, Grant SA. Anatomic evaluation of the sacral multifidus block. J Clin Anesth. 2021 Sep;72:110263. doi: 10.1016/j.jclinane.2021.110263. Epub 2021 Apr 5. No abstract available. PMID 33831768
- [Result] Ivanusic J, Konishi Y, Barrington MJ. A Cadaveric Study Investigating the Mechanism of Action of Erector Spinae Blockade. Reg Anesth Pain Med. 2018 Aug;43(6):567-571. doi: 10.1097/AAP.0000000000000789. PMID 29746445
- [Result] Aponte A, Sala-Blanch X, Prats-Galino A, Masdeu J, Moreno LA, Sermeus LA. Anatomical evaluation of the extent of spread in the erector spinae plane block: a cadaveric study. Can J Anaesth. 2019 Aug;66(8):886-893. doi: 10.1007/s12630-019-01399-4. Epub 2019 May 21. PMID 31119551
- [Derived] Keles BO, Salman N, Yilmaz ET, Birinci HR, Apan A, Ince S, Ozyasar AF, Uz A. Comparison of the median and intermediate approaches to the ultrasound-guided sacral erector spinae plane block: a cadaveric and radiologic study. Korean J Anesthesiol. 2024 Feb;77(1):156-163. doi: 10.4097/kja.23604. Epub 2023 Nov 15. PMID 37964515